CLINICAL TRIAL: NCT05373225
Title: Effect of Acetic Acid Shockwave Phonophoresis on Calcaneal Spur Patients: A Randomized Controlled Trial
Brief Title: Shockwave Phonophoresis on Calcaneal Spur Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Collaborators: Self (Unknown)
Responsible Party: Principal Investigator, Mostafa Ali Elwan, Assistance Lecturer at department of basic science and biomechanics at faculty of physical therapy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: shockwave phonophoresis
Record Dates: First submitted 2022-04-17; First posted 2022-05-13 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Calcaneal Spur
MeSH Terms: conditions — Heel Spur | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Shock wave Therapy (Experimental): This group will be composed of subjects who represented the experimental group 1. They will receive shock wave therapy
  Interventions: Device: Shock wave Therapy
- Acetic acid shockwave phonophoresis therapy (Experimental): This group will be composed of subjects who represented the experimental group 2. They will take 6 sessions with Time between sessions 5-7 days plus exercise and dietary advice
  Interventions: Device: Acetic acid shockwave phonophoresis therapy
- conventional physical therapy program (Active Comparator): This group will be composed of subjects who represented the control group
  Exercise program:
  * Standing calf-stretching exercise
  * Towel stretch: stretching exercise
  * Ice bottle
  * Towel pickup exercise
  * Marble pickups exercise
  * Calf raises exercises -Static and dynamic balance exercise
  Interventions: Other: conventional physical therapy program

INTERVENTIONS:
Device: Acetic acid shockwave phonophoresis therapy — This group composed of subjects. They will take 6 sessions with Time between sessions 5-7 days plus exercise and dietary advice
  Arms: Acetic acid shockwave phonophoresis therapy
Device: Shock wave Therapy — This group composed of subjects and represented the control group who will receive shock wave therapy
  Arms: Shock wave Therapy
Other: conventional physical therapy program — Exercise program:
  * Standing calf-stretching exercise
  * Towel stretch: stretching exercise
  * Ice bottle
  * Towel pickup exercise
  * Marble pickups exercise
  * Calf raises exercises -Static and dynamic balance exercise
  Arms: conventional physical therapy program

SUMMARY:
The Low energy shockwave has a significant effect on the permeability of tissue. Consequently, it might be used to deliver a substance such as Acetic acid. Accordingly, Shockwave might help to improve the outcomes with calcaneal spur patients. Therefore, the present study might help in the treatment of calcaneal spur patients and also might improve the quality of life in a fast and efficient way.

ELIGIBILITY:
Inclusion Criteria:

* Heel pain with a calcaneal spur.
* Calcaneal spur in a lateral calcaneal x-ray.
* Patient's age ranged from 30 to 65 years.
* Patients with a calcaneal spur.
* Patients with intact sensory perception.
* At least 6 weeks from last corticosteroid injection; 4 weeks from the last local anaesthetic injection, iontophoresis, ultrasound, and electrotherapy

Exclusion Criteria:

* History of fracture or surgery of the heel or ankle.
* Presence of inflammatory joint disease.
* Marked osteoporotic patient.
* Presence of ankylosing spondylitis or other inflammatory joint diseases.
* Heart pacemaker use.
* Patient on anticoagulant and coagulation disease.
* Skin wound or ulcers.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
calcaneal spur length by X-ray (mm) | three months
  X-ray on the affected foot to measure the length of the calcaneal spur
calcaneal spur width by X-ray (mm) | three months
  X-ray on the affected foot to measure the width of the calcaneal spur

SECONDARY OUTCOMES:
FPX 50 wagner Pressure pain threshold (PPT) | three months
  this device used to measure the pressure pain threshold
Activity of daily living: by Foot and Ankle Ability Measure scale | three months
  This scale formed from 29 item, the minimum score for each item is 0 and maximum score is 4 , the Higher scores represent higher levels of function for each subscale, with 100% representing no dysfunction
visual analogue scale. | three months
  this scale for pain intensity level assessment and contain minimum score is 0 and maximum score is 100 mm, the higher score indicate more pain (sever dysfunction)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT05373225/Prot_SAP_ICF_000.pdf